CLINICAL TRIAL: NCT01615003
Title: The Analysis of Blood Stasis Syndromeand of Coronary Heart Disease Related MicroRNA Genomics and Target Gene Regulatory Networks
Brief Title: The Study of MicroRNA Genomics of Blood Stasis Syndrome and of Coronary Heart Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNSF81173116
Record Dates: First submitted 2012-05-28; First posted 2012-06-08 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Heart Disease; Unstable Angina; Blood Stasis Syndrome
Keywords: MicroRNA; coronary heart disease; unstable angina; blood stasis syndrome; Xuesaitong soft capsule
MeSH Terms: conditions — Coronary Disease; Angina, Unstable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xuesaitong soft capsule group (Experimental): Patients who confirmed by coronary angiography and diagnosed blood stasis syndrome of coronary heart disease are given conventional Western medicine treatment and Xuesaitong soft capsule.
  Interventions: Drug: Xuesaitong soft capsule
- control group (Placebo Comparator): Patients who confirmed by coronary angiography and diagnosed blood stasis syndrome of coronary heart disease are given conventional Western medicine treatment and placebo.
  Interventions: Drug: Xuesaitong soft capsule Placebo

INTERVENTIONS:
Drug: Xuesaitong soft capsule — Xuesaitong soft capsule, soft capsule, Ingredients:PNS, Specification:0.33 per bag, once take two pills and twice a day during a month.
  Arms: Xuesaitong soft capsule group
Drug: Xuesaitong soft capsule Placebo — Xuesaitong soft capsule Placebo, soft capsule, once take two pills and twice a day during a month.
  Arms: control group

SUMMARY:
In this study, typical cases of blood stasis syndrome of coronary heart disease are selected, by using microRNA chip, cDNA microarray and other bioinformatics technologies to filter and verify related miRNA and its target gene of Coronary Heart disease. Meanwhile, intervene by Xuesaitong soft capsules to investigate related miRNA and its target gene of Coronary Heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coronary angiography unstable angina
* Clinical diagnosis of unstable angina
* Age of 30 to 75 years old
* Not use thrombolysis, dilate coronary drugs within two weeks
* Tongue dark
* Sign the consent

Exclusion Criteria:

* Severe valvular heart disease
* Insulin-dependent diabetes
* mental disease
* Combined with severe liver, kidney, hematopoietic system disorder
* Patients with malignant tumors
* Pregnancy or breast-feeding women
* Recent history of trauma
* Drug allergy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
the change of Cycle threshold of relational microRNA in coronary artery disease with unstable angina | 1 month
  The change of Cycle threshold of relational microRNA in coronary artery disease with unstable angina by real RT-PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'an men Hispital, Beijing, Beijing Municipality, China